CLINICAL TRIAL: NCT02004522
Title: A Phase 3 Study of Duvelisib Versus Ofatumumab in Patients With Relapsed or Refractory Chronic Lymphocytic Leukemia/ Small Lymphocytic Lymphoma (DUO)
Brief Title: A Phase 3 Study of Duvelisib Versus Ofatumumab in Patients With Relapsed or Refractory CLL/SLL (DUO)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SecuraBio (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IPI-145-07; 2013-002405-61 (EudraCT Number)
Record Dates: First submitted 2013-11-13; First posted 2013-12-09 (Estimated); Results first posted 2019-01-08 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma
Keywords: Phase 3; CLL/SLL; Pi3K
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — duvelisib; ofatumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Duvelisib (Experimental): Duvelisib is administered orally and supplied as 5 mg and 25 mg formulated capsules.
  Interventions: Drug: Duvelisib
- Ofatumumab (Active Comparator): Ofatumumab is administered as an intravenous (IV) infusion and is supplied in single-use vials at two strengths, 100 mg/5 mL and 1000 mg/50 mL.
  Interventions: Drug: Ofatumumab

INTERVENTIONS:
Drug: Duvelisib — PI3K Inhibitor
  Other Names: Copiktra, IPI-145, PI3K Inhibitor
  Arms: Duvelisib
Drug: Ofatumumab — monoclonal antibody
  Other Names: Arzerra
  Arms: Ofatumumab

SUMMARY:
A Phase 3 clinical trial to examine the efficacy of duvelisib monotherapy versus ofatumumab monotherapy in subjects with relapsed or refractory Chronic Lymphocytic Leukemia (CLL) or Small Lymphocytic Lymphoma (SLL).

DETAILED DESCRIPTION:
This is an open-label, two- arm, randomized phase 3, superiority trial designed to evaluate the efficacy and safety of duvelisib compared to ofatumumab administered to patients who have been diagnosed with CLL/SLL whose disease is relapsed or refractory.

Approximately 150 subjects will receive a starting dose of 25 mg duvelisib BID initially over the course of 21-day treatment cycle followed by 28-day treatment cycles for up to 18 cycles or until disease progression or unacceptable toxicity (whichever comes first). After 18 complete cycles of treatment, subjects may receive additional cycles of duvelisib until disease progression or unacceptable toxicity if they, in the judgment of the Investigator, may derive benefit from continued treatment, and if the subject meets the criteria for additional treatment at Cycle 19 Day 1.

Approximately 150 subjects will receive a starting dose of 300 mg ofatumumab on Day 1 followed by seven weekly doses of 2000 mg. Thereafter, subjects will receive 2000 mg ofatumumab once every month for four months. Administration of ofatumumab will not exceed the 12 doses (within 7 cycles).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of active CLL or SLL that meets at least one of the IWCLL 2008 criteria for requiring treatment (Binet Stage ≥ B and/or Rai Stage ≥ I)
* Disease that has progressed during or relapsed after at least one previous CLL/SLL therapy
* Not appropriate for treatment with a purine-based analogue regimen (per National Comprehensive Cancer Network [NCCN] or European Society for Medical Oncology [ESMO] guidelines), including relapse ≤ 36 months from a purine-based chemoimmunotherapy regimen or relapse ≤ 24 months from a purine-based monotherapy regimen
* A cytogenetics or fluorescence in situ hybridization (FISH) analysis of the leukemic cells within 24 months of randomization is required to document the presence or absence of del(17p). Note: if a sample from within 24 months is not available, it should be evaluated as part of the screening laboratory evaluation to inform stratification
* Measurable disease with a lymph node or tumor mass > 1.5 cm in at least one dimension as assessed by computed tomography (CT)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2 (corresponds to Karnofsky Performance Status [KPS] ≥ 60%)
* Willingness by subject to be randomized to receive either ofatumumab or duvelisib at the dose and schedule defined in the protocol
* Must meet the following laboratory parameters:

  1. Serum aspartate transaminase (AST/SGOT) or alanine transaminase (ALT/SGPT) ≤ 3 x upper limit of normal (ULN)
  2. Total bilirubin ≤ 1.5 x ULN
  3. Serum creatinine ≤ 2.0 x ULN
  4. Hemoglobin ≥ 8.0 g/dL with or without transfusion support
  5. Platelet count ≥ 10,000 μL with or without transfusion support
* For women of childbearing potential (WCBP): negative serum β-human chorionic gonadotropin (βhCG) pregnancy test within 1 week before randomization (WCBP defined as a sexually mature woman who has not undergone surgical sterilization or who has not been naturally post-menopausal for at least 24 consecutive months [women ≤ 55 years] or 12 consecutive months [women > 55 years])
* Willingness of male and female subjects who are not surgically sterile or postmenopausal to use medically acceptable methods of birth control from the first dose of study drug to 30 days after the last dose of duvelisib and for 12 months after last dose of ofatumumab. Sexually active men, and women using oral contraceptive pills, should also use barrier contraception
* Ability to voluntarily sign consent for and adhere to the entire study visit schedule and all protocol requirements
* Signed and dated institutional review board (IRB)/independent ethics committee (IEC)-approved informed consent form (ICF) before any study specific screening procedures are performed

Exclusion Criteria:

* History of Richter's transformation or prolymphocytic leukemia
* Uncontrolled autoimmune hemolytic anemia (AIHA) or idiopathic thrombocytopenia purpura (ITP) that is uncontrolled or requiring > 20 mg once daily (QD) of prednisone (or equivalent) to maintain hemoglobin > 8.0 g/dL or platelets > 10,000 μL without transfusion support
* Refractory to ofatumumab (progression or relapse <12 months of receiving ofatumumab therapy or <24 months of receiving an ofatumumab- containing regimen)
* Prior allogeneic transplant (prior autologous stem cell transplant >6 months prior to study entry is permitted)
* Known central nervous system lymphoma or leukemia; subjects with symptoms of CNS disease must have a negative CT scan or negative diagnostic lumbar puncture prior to randomization
* Use of any of the following medications or procedures within the specified timeframe:
* Use of live or live attenuated vaccines within 30 days prior to randomization
* Chemotherapy, radiation therapy, or ablative therapy within 3 weeks of randomization
* Tyrosine kinase inhibitor within 7 days of randomization
* Other investigational therapy (not included above) within 3 weeks of randomization
* Previous treatment with a PI3K inhibitor or BTK inhibitor
* Ongoing treatment with chronic immunosuppressants (eg, cyclosporine) or systemic steroids > 20 mg prednisone (or equivalent) QD
* History of tuberculosis treatment within the preceding two years
* Ongoing systemic bacterial, fungal, or viral infections at the time of initiation of study treatment (defined as requiring IV antimicrobial, antifungal or antiviral agents)
* Subjects on antimicrobial, antifungal or antiviral prophylaxis are not specifically excluded if all other inclusion/exclusion criteria are met and there is no evidence of active infection at randomization
* Human immunodeficiency virus (HIV) infection
* Prior, current, or chronic hepatitis B or hepatitis C infection
* History of alcohol abuse or chronic liver disease (other than metastatic disease to the liver)
* Unable to receive prophylactic treatment for pneumocystis or herpes simplex virus (HSV)
* Baseline QT interval corrected with Fridericia's method (QTcF) > 480 ms (average of triplicate readings) Note: This criterion does not apply to subjects with a right or left bundle branch block (BBB)
* Unstable or severe uncontrolled medical condition (eg, unstable cardiac function, unstable pulmonary condition), or any important medical illness or abnormal laboratory finding that would, in the investigator's judgment, increase the subject's risk while participating in this study
* Concurrent active malignancy other than nonmelanoma skin cancer or carcinoma in situ of the cervix, bladder, or prostate not requiring treatment. Subjects with previous malignancies are eligible provided that they have been disease free for ≥2 years
* History of stroke, unstable angina, myocardial infarction, or ventricular arrhythmia requiring medication or mechanical control within the last 6 months
* Administration of medications or foods that are strong inhibitors or inducers of CYP3A within 2 weeks of randomization
* Prior surgery or gastrointestinal dysfunction that may affect drug absorption (eg, gastric bypass surgery, gastrectomy)
* Major surgery or invasive intervention within 4 weeks prior to randomization
* Pregnant or breastfeeding women
* Hypersensitivity to ofatumumab or its excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 319 (Actual)
Dates: Start 2013-11; Primary Completion 2017-05-19 (Actual); Study Completion 2021-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (83):
- United States (35):
  - La Jolla, California
  - Denver, Colorado
  - Altamonte Springs, Florida
  - Bonita Springs, Florida
  - Bradenton, Florida
  - Brandon, Florida
  - Cape Coral, Florida
  - Clearwater, Florida
  - Englewood, Florida
  - Fort Myers, Florida
  - Gainesville, Florida
  - Hudson, Florida
  - Inverness, Florida
  - Largo, Florida
  - Naples, Florida
  - New Port Richey, Florida
  - Orange City, Florida
  - Orlando, Florida
  - Port Charlotte, Florida
  - Sarasota, Florida
  - Spring Hill, Florida
  - St. Petersburg, Florida
  - Tampa, Florida
  - Tavares, Florida
  - Venice, Florida
  - Crestview Hills, Kentucky
  - Boston, Massachusetts
  - St Louis, Missouri
  - Hackensack, New Jersey
  - New Brunswick, New Jersey
  - New York, New York
  - Cincinnati, Ohio
  - Fairfield, Ohio
  - Nashville, Tennessee
  - Charlottesville, Virginia
- Australia (3):
  - Bedford Park
  - East Melbourne
  - Melbourne
- Austria (2):
  - Vienna
  - Wels
- Belgium (4):
  - Brussels
  - Ghent
  - Leuven
  - Sint-Niklaas
- France (10):
  - Argenteuil
  - Bobigny
  - Bordeaux
  - Caen
  - Clermont-Ferrand
  - La Roche-sur-Yon
  - Limoges
  - Nantes
  - Rennes
  - Vendœuvres
- Germany (5):
  - Berlin
  - Cologne
  - Leer
  - Rostock
  - Ulm
- Hungary (6):
  - Budapest
  - Debrecen
  - Győr
  - Kaposvár
  - Pécs
  - Szeged
- Italy (8):
  - Catania
  - Lecce
  - Meldola
  - Milan
  - Padua
  - Ravenna
  - Rimini
  - Roma
- New Zealand (2):
  - Auckland
  - Palmerston North
- Spain (3):
  - Barcelona
  - Madrid
  - Pamplona
- United Kingdom (5):
  - Bournemouth
  - Leeds
  - Manchester
  - Nottingham
  - Oxford

REFERENCES:
- [Derived] Flinn IW, Hillmen P, Montillo M, Nagy Z, Illes A, Etienne G, Delgado J, Kuss BJ, Tam CS, Gasztonyi Z, Offner F, Lunin S, Bosch F, Davids MS, Lamanna N, Jaeger U, Ghia P, Cymbalista F, Portell CA, Skarbnik AP, Cashen AF, Weaver DT, Kelly VM, Turnbull B, Stilgenbauer S. The phase 3 DUO trial: duvelisib vs ofatumumab in relapsed and refractory CLL/SLL. Blood. 2018 Dec 6;132(23):2446-2455. doi: 10.1182/blood-2018-05-850461. Epub 2018 Oct 4. PMID 30287523

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Duvelisib | Ofatumumab
Started (Number of subjects randomized.) | 160 | 159
Number of Subjects Treated (Number of subjects exposed to treatment.) | 158 | 155
Completed | 34 (Completed defined here as still on treatment.) | 0 (Completed defined here as still on treatment.)
Not Completed | 126 | 159
Not completed — Adverse Event | 55 | 6
Not completed — Withdrawal by Subject | 13 | 7
Not completed — Death | 12 | 3
Not completed — Physician Decision | 3 | 4
Not completed — Protocol Violation | 1 | 0
Not completed — Other is reason listed by PI | 4 | 1
Not completed — Never Dosed | 2 | 4
Not completed — Disease Progression | 35 | 31
Not completed — Completed Treatment Cycles Per Protocol | 1 | 103

BASELINE CHARACTERISTICS:
Groups:
- Ofatumumab: Ofatumumab is administered as an IV infusion and is supplied in single-use vials at two strengths, 100 mg/5 mL and 1000 mg/50 mL.
- Total: Total of all reporting groups
Arm/Group | Duvelisib | Ofatumumab | Total
Number analyzed (Participants) | 160 | 159 | 319
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 48 | 54 | 102
  >=65 years | 112 | 105 | 217
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 64 | 128
  Male | 96 | 95 | 191
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 7 | 15
  Not Hispanic or Latino | 130 | 133 | 263
  Unknown or Not Reported | 22 | 19 | 41
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 150 | 142 | 292
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 9 | 16 | 25
Region of Enrollment [Number; unit: participants]
  New Zealand | 6 | 6 | 12
  Austria | 3 | 8 | 11
  Belgium | 13 | 14 | 27
  Hungary | 35 | 30 | 65
  United States | 30 | 21 | 51
  Italy | 23 | 18 | 41
  United Kingdom | 7 | 10 | 17
  Australia | 9 | 12 | 21
  France | 12 | 18 | 30
  Germany | 1 | 3 | 4
  Spain | 21 | 19 | 40

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: The primary efficacy endpoint for the study was PFS, defined as time from randomization to the first documentation of PD as determined by blinded independent review or death due to any cause.
Time Frame: From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 3 years
Population: Intent to Treat
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Duvelisib | Ofatumumab
Number analyzed (Participants) | 160 | 159
Months | 13.3 [12.1 to 16.8] | 9.9 [9.2 to 11.3]

2. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR is a key secondary efficacy endpoint with overall response defined as best response of CR, CRi, PR, or PRwL, according to the modified IWCLL/IWG Response Criteria, with modification for treatment-related lymphocytosis as defined in the protocol.
Time Frame: Until disease progression or unacceptable toxicity assessed up to 6 years
Population: Intent to Treat
Measure: Count of Participants; unit: Participants
Arm/Group | Duvelisib | Ofatumumab
Number analyzed (Participants) | 160 | 159
Participants | 118 | 72

3. Secondary Outcome: Number of Subjects With Hematologic Improvements
Description: Subjects with hematologic improvement included those subjects with abnormally high values for neutrophil count, hemoglobin, or platelet count at Baseline determined to have consistently met the criteria of an improvement for those parameters for a period of at least 60 days during which the subject did not have a transfusion or exogenous cytokines.
Time Frame: 3 years
Population: Subjects With Abnormal Hematologic Values at Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Duvelisib | Ofatumumab
Number analyzed (Participants) | 94 | 95
Participants | 56 | 51

4. Secondary Outcome: Overall Survival
Description: A stratified Cox regression analysis was used to test for any treatment effect.
Time Frame: Every 6 months for up to 3 years after first dose
Population: Intent to Treat
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Duvelisib | Ofatumumab
Number analyzed (Participants) | 160 | 159
Months | 54.94 [43.00 to 67.99] | 63.25 [44.15 to NA] — NA = The upper limit of the confidence interval is not estimable because of an insufficient number of events at the time of analysis.

5. Secondary Outcome: Lymph Node Response Rate
Description: Lymph node response defined as greater than or equal to 50% decrease in the SPD of target lymph nodes
Time Frame: 3 years
Population: Intent to Treat
Measure: Count of Participants; unit: Participants
Arm/Group | Duvelisib | Ofatumumab
Number analyzed (Participants) | 160 | 159
Participants | 136 | 25

6. Secondary Outcome: Duration of Response (DOR)
Description: Duration of response is defined only for subjects demonstrating a response (eg, CR, CRi, PR, PRwL), with the response and progression statuses both determined by the blinded, central independent review. The analysis will be descriptive for each treatment group only.
Time Frame: Time from the first documentation of response to first documentation of progressive disease or death due to any cause
Population: Intent to Treat
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Duvelisib | Ofatumumab
Number analyzed (Participants) | 160 | 159
Months | 11.1 [9.2 to 18.3] | 9.3 [7.7 to 11.0]

7. Secondary Outcome: Treatment-Emergent Adverse Events (TEAEs) and Changes in Safety Laboratory Values
Description: An analysis of TEAEs with an onset within the first 24 weeks of treatment was performed to examine and compare the incidence of events across an equal period for each treatment arm.Twenty-four weeks was anticipated to be the median exposure to ofatumumab.
Time Frame: From 04 Feb 2014 till 19 June 2018
Population: Intent to Treat
Measure: Count of Participants; unit: Participants
Arm/Group | Duvelisib | Ofatumumab
Number analyzed (Participants) | 160 | 159
Participants | 150 | 143

8. Secondary Outcome: Number of Subjects With Samples Available for Duvelisib Pharmacokinetics (PK)
Description: Number of subjects with samples available for duvelisib Pharmacokinetics (PK)
Time Frame: Cycle 2, Cycle 3, and Cycle 7
Population: Intent to Treat for duvelisib patients, no PK samples were collected for ofatumumab patients.
Measure: Number; unit: participants
Arm/Group | Duvelisib
Number analyzed (Participants) | 160
participants | 158

ADVERSE EVENTS:
Time Frame: 39 months
Description: Safety data rerun to include treatment-emergent adverse events that occurred on Day 1.
Arm/Group | Duvelisib | Ofatumumab
All-Cause Mortality (participants affected / at risk) | 78/158 | 70/155
Serious Adverse Events (participants affected / at risk) | 124/158 | 50/155
Other Adverse Events (participants affected / at risk) | 149/158 | 130/155
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Duvelisib (N=158) | Ofatumumab (N=155)
Febrile neutropenia (Blood and lymphatic system disorders) | 10 | 3
Anaemia (Blood and lymphatic system disorders) | 2 | 2
Haemolytic anaemia (Blood and lymphatic system disorders) | 2 | 1
Pancytopenia (Blood and lymphatic system disorders) | 3 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Lymph node pain (Blood and lymphatic system disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 2 | 1
Cardiac failure (Cardiac disorders) | 3 | 1
Cardiac failure congestive (Cardiac disorders) | 2 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Pericarditis (Cardiac disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 20 | 1
Diarrhoea (Gastrointestinal disorders) | 18 | 1
Enterocolitis (Gastrointestinal disorders) | 2 | 1
Gastritis (Gastrointestinal disorders) | 3 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Colitis ischaemic (Gastrointestinal disorders) | 1 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0
Mallory-Weiss syndrome (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Proctitis (Gastrointestinal disorders) | 1 | 0
Oesophageal ulcer (Gastrointestinal disorders) | 0 | 1
Portal hypertensive gastropathy (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Ileal ulcer (Gastrointestinal disorders) | 1 | 0
Death (General disorders) | 2 | 0
Mucosal inflammation (General disorders) | 1 | 0
Multi-organ failure (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Sudden death (General disorders) | 1 | 0
Disease progression (General disorders) | 0 | 2
Fatigue (General disorders) | 0 | 1
Infusion site extravasation (General disorders) | 0 | 1
Pyrexia (General disorders) | 7 | 1
General physical health deterioration (General disorders) | 4 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 1
Contrast media allergy (Immune system disorders) | 0 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 1
Pneumocystis jirovecii pneumonia (Infections and infestations) | 3 | 0
Pneumonia pneumococcal (Infections and infestations) | 3 | 0
Pneumonia pseudomonas aeruginosa (Infections and infestations) | 3 | 0
Sepsis (Infections and infestations) | 3 | 1
Upper respiratory tract infection (Infections and infestations) | 3 | 0
Aspergillus infection (Infections and infestations) | 2 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 2 | 0
Campylobacter gastroenteritis (Infections and infestations) | 2 | 0
Clostridium difficile colitis (Infections and infestations) | 2 | 0
Fungal infection (Infections and infestations) | 2 | 0
Influenza (Infections and infestations) | 2 | 0
Lower respiratory tract infection (Infections and infestations) | 2 | 1
Pneumonia bacterial (Infections and infestations) | 2 | 2
Pneumonia staphylococcal (Infections and infestations) | 2 | 0
Pseudomonal sepsis (Infections and infestations) | 2 | 0
Skin infection (Infections and infestations) | 2 | 0
Urinary tract infection (Infections and infestations) | 2 | 0
Bronchiolitis (Infections and infestations) | 1 | 0
Bronchitis viral (Infections and infestations) | 1 | 0
Bronchopneumonia (Infections and infestations) | 1 | 0
Cytomegalovirus colitis (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0
Enterococcal infection (Infections and infestations) | 1 | 0
Enterococcal sepsis (Infections and infestations) | 1 | 0
Escherichia sepsis (Infections and infestations) | 1 | 3
Escherichia urinary tract infection (Infections and infestations) | 1 | 2
Gastroenteritis viral (Infections and infestations) | 1 | 0
Haemophilus infection (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 0
Infusion site cellulitis (Infections and infestations) | 1 | 0
Lobar pneumonia (Infections and infestations) | 1 | 0
Lower respiratory tract infection viral (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 1 | 0
Pneumonia escherichia (Infections and infestations) | 1 | 0
Pneumonia klebsiella (Infections and infestations) | 1 | 0
Pneumonia mycoplasmal (Infections and infestations) | 1 | 0
Pneumonia respiratory syncytial viral (Infections and infestations) | 1 | 0
Pneumonia streptococcal (Infections and infestations) | 1 | 0
Pseudomonas bronchitis (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0
Respiratory tract infection bacterial (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 1 | 0
Streptococcal bacteraemia (Infections and infestations) | 1 | 1
Streptococcal sepsis (Infections and infestations) | 1 | 0
Wound infection staphylococcal (Infections and infestations) | 1 | 0
Chronic sinusitis (Infections and infestations) | 0 | 1
Clostridium difficile infection (Infections and infestations) | 0 | 1
Device related infection (Infections and infestations) | 0 | 1
Herpes virus infection (Infections and infestations) | 0 | 1
Pneumonia viral (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 4 | 1
Pneumonia (Infections and infestations) | 25 | 5
Bronchitis (Infections and infestations) | 5 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Splenic rupture (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 3
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Lipase increased (Investigations) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1
Malnutrition (Metabolism and nutrition disorders) | 1 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Intestinal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Neuroendocrine carcinoma of the skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Haemorrhagic stroke (Nervous system disorders) | 2 | 0
Brain stem haemorrhage (Nervous system disorders) | 1 | 0
Dementia (Nervous system disorders) | 1 | 0
Mental impairment (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Renal colic (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Renal failure chronic (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 4 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Laryngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 6 | 0
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 2 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 4 | 0
Deep vein thrombosis (Vascular disorders) | 2 | 1
Hypertension (Vascular disorders) | 1 | 0
Thrombosis (Vascular disorders) | 1 | 0
Peripheral embolism (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Duvelisib (N=158) | Ofatumumab (N=155)
Neutropenia (Blood and lymphatic system disorders) | 53 | 32
Anaemia (Blood and lymphatic system disorders) | 39 | 16
Thrombocytopenia (Blood and lymphatic system disorders) | 27 | 9
Diarrhoea (Gastrointestinal disorders) | 79 | 19
Nausea (Gastrointestinal disorders) | 38 | 17
Constipation (Gastrointestinal disorders) | 27 | 12
Vomiting (Gastrointestinal disorders) | 23 | 10
Abdominal pain (Gastrointestinal disorders) | 17 | 3
Dyspepsia (Gastrointestinal disorders) | 9 | 4
Abdominal pain upper (Gastrointestinal disorders) | 9 | 5
Paraesthesia oral (Gastrointestinal disorders) | 0 | 10
Colitis (Gastrointestinal disorders) | 8 | 1
Dry mouth (Gastrointestinal disorders) | 8 | 1
Pyrexia (General disorders) | 46 | 15
Fatigue (General disorders) | 25 | 18
Asthenia (General disorders) | 20 | 17
Oedema peripheral (General disorders) | 16 | 7
Pneumonia (Infections and infestations) | 8 | 4
Bronchitis (Infections and infestations) | 20 | 12
Upper respiratory tract infection (Infections and infestations) | 22 | 12
Nasopharyngitis (Infections and infestations) | 13 | 4
Respiratory tract infection (Infections and infestations) | 11 | 3
Infusion related reaction (Injury, poisoning and procedural complications) | 2 | 28
Alanine aminotransferase increased (Investigations) | 13 | 3
Weight decreased (Investigations) | 21 | 3
Aspartate aminotransferase increased (Investigations) | 15 | 3
Dehydration (Metabolism and nutrition disorders) | 8 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 16 | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 11 | 5
Decreased appetite (Metabolism and nutrition disorders) | 24 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 12 | 8
Muscle spasms (Musculoskeletal and connective tissue disorders) | 7 | 8
Dizziness (Nervous system disorders) | 13 | 5
Headache (Nervous system disorders) | 13 | 13
Paraesthesia (Nervous system disorders) | 7 | 15
Insomnia (Psychiatric disorders) | 8 | 9
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 9 | 3
Productive cough (Respiratory, thoracic and mediastinal disorders) | 8 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 36 | 22
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 14 | 9
Rash (Skin and subcutaneous tissue disorders) | 17 | 18
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 9 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 11 | 9
Hypertension (Vascular disorders) | 13 | 4
Hypotension (Vascular disorders) | 4 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-02-09): https://cdn.clinicaltrials.gov/large-docs/22/NCT02004522/Prot_001.pdf
  • Statistical Analysis Plan (2017-05-09): https://cdn.clinicaltrials.gov/large-docs/22/NCT02004522/SAP_000.pdf